CLINICAL TRIAL: NCT05425524
Title: Leptospirosis Care Bundle Study: A Randomized Controlled Trial
Brief Title: Leptospirosis Care Bundle Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Assoc. Prof. Dr.Nattachai Srisawat, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB.521/62
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Leptospirosis
MeSH Terms: conditions — Leptospirosis | interventions — Patient Care Bundles

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care Bundle Group (Experimental): Treatment step by step we have 5 steps STEP 1: Leptospirosis suspected case STEP 2: Investigations STEP 3: Antibiotics within 1 hour after Hemocultures were taken STEP 4: Intravenous Fluid STEP 5: Stage-Base Management of AKI (KDIGO)
  Interventions: Procedure: Care Bundle
- Control Group (No Intervention)

INTERVENTIONS:
Procedure: Care Bundle — Treatment step by step we have 5 steps STEP 1: Leptospirosis suspected case STEP 2: Investigations STEP 3: Antibiotics within 1 hour after Hemocultures were taken STEP 4: Intravenous Fluid STEP 5: Stage-Base Management of AKI (KDIGO)
  Arms: Care Bundle Group

SUMMARY:
So in management of Leptospirosis patients There really is no another approach to treatment. The importance of the problem was acknowledged by the researchers. As a result, this study was performed in order to The Leptospirosis Care Bundle has been used, and has been proved that its use can reduce the risk of acute renal failure.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Suspicious Leptospirosis including body temperature > 38 celcius, Severe myalgia, and exposure to reservoir hospital of flood water.
* Calf muscle tenderness
* Conjunctival suffusion
* Anuria or oliguria and/or proteinuria
* Jaundice
* Hemorrhagic manifestations (pulmonary and intestine)
* Meningeal irritation
* Nausea, vomiting, abdominal pain, diarrhea.
* Admitted in hospital

Exclusion Criteria:

* other infectious disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Reduce AKI in 72 hours | 72 hours
  To see if using care bundle for leptospirosis patients can improve reduce the incidence of acute renal failure in the first 72 hours of being admitted to hospital.It classified AKI into three categories (risk, injury, and failure) according to the status of serum creatinine (SCr) and urine output (UO) by AKIN/KDIGO

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn university, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No